CLINICAL TRIAL: NCT01213316
Title: A Non-interventional Cohort Study for the Assessment of the Efficacy of RALTEGRAVIR 400 mg Administered Twice Daily in Combination With Other Antiretroviral Drugs to Treat Infection With the Human Immunodeficiency Virus 1 (HIV-1) in Adults and Aging Patients (≥ 50 Years) Under Conditions That Are Representative of the Nationwide Treatment of HIV-positive Patients in Germany
Brief Title: A Study to Assess the Efficacy of Raltegravir (Isentress®), Administered in Combination With Other Antiretroviral Drugs as Treatment for Adults and Older Adults Infected With the Human Immunodeficiency Virus 1 (HIV-1)(MK-0518-145) (Wirksamkeit Von Isentress® Unter Praxisbedingungen)
Acronym: WIP
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0518-145
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: HIV-1 Infection
Keywords: HIV; antiretroviral; human immunodeficiency virus; Raltegravir; Adults with HIV-1 infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Overall Participants: HIV-1 infected participants received raltegravir 400 mg tablet orally twice daily for 96 weeks (Initial Cohort), 144 weeks (Prolonged Cohort) or 48 weeks (Amendment Cohort) in combination with other antiretroviral drugs under conditions representative of standard of clinical practice for HIV-1 patients in Germany.
  Interventions: Drug: Raltegravir
- Aging Participants: HIV-1 infected participants received raltegravir 400 mg tablet orally twice daily for 144 weeks (Prolonged Cohort) or 48 weeks (Amendment Cohort) in combination with other antiretroviral drugs under conditions representative of standard of clinical practice for HIV-1 patients in Germany.
  Includes newly enrolled participants ≥ 50 years of age (Amendment Cohort), plus participants from the Initial Cohort who were ≥ 50 years of age at time of recruitment and who completed 48 weeks of treatment (Prolonged Cohort).
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Raltegravir, 400 mg, per oral (p.o.) twice daily (b.i.d.) for 48 or 144 weeks
  Other Names: ISENTRESS®
  Groups: Aging Participants
Drug: Raltegravir — Raltegravir, 400 mg, per oral (p.o.) twice daily (b.i.d.) for 96, 144, or 48 weeks
  Other Names: ISENTRESS®
  Groups: Overall Participants

SUMMARY:
This is an observational, non-comparative, multicenter, open-label study. Participants will be treated with Raltegravir according to standard clinical practice, and monitored over a total period of 96 weeks. In an extension to the study (Amendment 1), a new cohort of aging participants (≥ 50 years) will be recruited and monitored over a total period of 48 weeks. Participants who stop taking Raltegravir before the end of the 96-week period or 48-week period, respectively, will be followed up for 3 months after discontinuing the drug. The primary objective is to determine the proportion of participants with a human immunodeficiency virus (HIV)-1 viral load < 50 copies/mL after 48 weeks of treatment with Raltegravir.

ELIGIBILITY:
Inclusion Criteria

The prospective participant must meet, at least, all of the criteria below to be eligible for study participation. The participant:

* Is a minimum age of 18 years (adults) or 50 years (aging participants);
* Is male or female;
* Has confirmed infection with HIV-1 (positive HIV test according to appropriate standard practice);
* Has commenced antiretroviral treatment with Raltegravir according to the recommendations made in the Summary of Product Characteristics at the time of enrollment on the study, or a maximum 6 months prior to enrollment on the study;
* Has any cluster of differentiation (CD4) cell (specialized white blood cell) count upon enrollment on the study.

Exclusion criteria

If the prospective participant meets any of the criteria below (among others determined by the study staff) they will NOT be eligible for study participation. The participant:

* For which Raltegravir, or its ingredients, are contraindicated;
* Has intolerance to Raltegravir, or its ingredients;
* If female, is pregnant, breastfeeding, or is planning a pregnancy or egg donation during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with confirmed HIV-1 infection
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2010-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Friis-Moller N, Thiebaut R, Reiss P, Weber R, Monforte AD, De Wit S, El-Sadr W, Fontas E, Worm S, Kirk O, Phillips A, Sabin CA, Lundgren JD, Law MG; DAD study group. Predicting the risk of cardiovascular disease in HIV-infected patients: the data collection on adverse effects of anti-HIV drugs study. Eur J Cardiovasc Prev Rehabil. 2010 Oct;17(5):491-501. doi: 10.1097/HJR.0b013e328336a150. PMID 20543702
- [Background] D'Agostino RB Sr, Vasan RS, Pencina MJ, Wolf PA, Cobain M, Massaro JM, Kannel WB. General cardiovascular risk profile for use in primary care: the Framingham Heart Study. Circulation. 2008 Feb 12;117(6):743-53. doi: 10.1161/CIRCULATIONAHA.107.699579. Epub 2008 Jan 22. PMID 18212285
- [Background] Anderson KM, Odell PM, Wilson PW, Kannel WB. Cardiovascular disease risk profiles. Am Heart J. 1991 Jan;121(1 Pt 2):293-8. doi: 10.1016/0002-8703(91)90861-b. PMID 1985385
- [Background] Anderson KM, Wilson PW, Odell PM, Kannel WB. An updated coronary risk profile. A statement for health professionals. Circulation. 1991 Jan;83(1):356-62. doi: 10.1161/01.cir.83.1.356. No abstract available. PMID 1984895
- [Derived] Naumann U, Moll A, Schleehauf D, Lutz T, Schmidt W, Jaeger H, Funke B, Witte V. Similar efficacy and tolerability of raltegravir-based antiretroviral therapy in HIV-infected patients, irrespective of age group, burden of comorbidities and concomitant medication: Real-life analysis of the German 'WIP' cohort. Int J STD AIDS. 2017 Aug;28(9):893-901. doi: 10.1177/0956462416679550. Epub 2016 Nov 14. PMID 28385065

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Initial Cohort included participants >=18 years old to receive treatment for 96 weeks. With the amendment, participants in the initial cohort >=50 years old could continue for an additional 48-weeks observation (Prolonged Cohort), and participants >=50 years old were newly enrolled to receive treatment for 48 weeks (Amendment Cohort).
Period: Overall Study
Arm/Group | Overall Participants
Started | 451 (Participants in the initial and amendment cohorts)
Amendment Cohort: Prolonged Participants | 48 (Participants >=50 years of age in the initial cohort who accept an additional 48-week observation)
Amendment Cohort: Newly Enrolled | 179 (Participants >=50 years of age newly enrolled)
Discontinued Treatment Before 48 Weeks | 67
Initial Cohort | 272 (Participants >=18 years of age in the initial cohort)
Completed | 451
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Participants
Number analyzed (Participants) | 451
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 382

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an HIV-1 Viral Load <50 Copies/mL After 48 Weeks of Raltegravir Treatment
Description: The percentage of participants with an HIV-1 viral load <50 copies/mL of HIV-1 RNA after 48 weeks of raltegravir treatment was determined.
Time Frame: Baseline and 48 weeks
Population: The analysis set included all participants who received at least one dose of raltegravir during the observation period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Overall Participants
Number analyzed (Participants) | 451
Percentage of participants
  Baseline | 50.8 [46.1 to 55.5]
  48 weeks | 74.7 [70.4 to 78.7]

2. Primary Outcome: Percentage of Aging Participants With an HIV-1 Viral Load <50 Copies/mL After 48 Weeks of Raltegravir Treatment
Description: The percentage of aging participants (>=50 years old at initiation of raltegravir treatment) with an HIV-1 viral load <50 copies/mL of HIV-1 RNA after 48 weeks of raltegravir treatment was determined.
Time Frame: Baseline and 48 weeks
Population: The analysis set included aging participants (Prolonged Participants and Newly Enrolled Participants) who received at least one dose of raltegravir during the observation period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Aging Participants: HIV-1 infected participants >=50 years old received raltegravir 400 mg tablet orally twice daily for 144 weeks (Prolonged Cohort) or 48 weeks (Amendment Cohort) in combination with other antiretroviral drugs under conditions representative of standard of clinical practice for HIV-1 patients in Germany.
Arm/Group | Aging Participants
Number analyzed (Participants) | 227
Percentage of participants
  Baseline | 62.1 [55.5 to 68.4]
  48 weeks | 77.5 [71.5 to 82.8]

3. Secondary Outcome: Percentage of Participants With an HIV-1 Viral Load <50 Copies/mL After 96 Weeks of Raltegravir Treatment
Description: The percentage of participants with an HIV-1 viral load <50 copies/mL of HIV-1 RNA after 96 weeks of raltegravir treatment was determined.
Time Frame: Baseline and 96 weeks
Population: The analysis set included participants in the Initial Cohort who received at least one dose of raltegravir during the observation period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Initial Cohort Participants: HIV-1 infected participants received raltegravir 400 mg tablet orally twice daily for 96 weeks in combination with other antiretroviral drugs under conditions representative of standard clinical practice for HIV-1 patients in Germany.
Arm/Group | Initial Cohort Participants
Number analyzed (Participants) | 272
Percentage of participants
  Baseline | 43.8 [37.8 to 49.9]
  96 weeks | 68.0 [62.1 to 73.5]

4. Secondary Outcome: HIV-1 Viral Load After 96 Weeks of Raltegravir Treatment
Description: The HIV-1 viral load (log10 copies/mL of HIV-1 RNA) was determined at Baseline and after 96 weeks of raltegravir treatment.
Time Frame: Baseline and 96 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Log10 Copies/mL
Arm/Group | Initial Cohort Participants
Number analyzed (Participants) | 272
Log10 Copies/mL
  Baseline | 2.90 (1.65) [62.1 to 73.5]
  96 weeks | 1.52 (0.43)

5. Secondary Outcome: Change From Baseline in CD4+ T-cell Counts After 96 Weeks of Raltegravir Treatment
Description: Mean CD4+ T-cell counts were determined at baseline and after 96 weeks of raltegravir treatment. A positive change from baseline indicates an increase in CD4+ T-cell count.
Time Frame: Baseline and 96 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: CD4+ T-cells/µL
Arm/Group | Initial Cohort Participants
Number analyzed (Participants) | 272
CD4+ T-cells/µL
  Baseline | 461.9 (286.35) [131.4 to 192.1]
  Change from Baseline at 96 weeks: n=216 | 161.7 (225.98) [131.4 to 192.1]

6. Secondary Outcome: HIV-1 Viral Load in Aging Participants After 48 Weeks of Raltegravir Treatment
Description: The HIV-1 viral load (log10 copies/mL of HIV-1 RNA) was determined in aging participants (>=50 years old at initiation of raltegravir treatment) at Baseline and after 48 weeks of raltegravir treatment.
Time Frame: Baseline and 48 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 Copies/mL
Arm/Group | Aging Participants
Number analyzed (Participants) | 227
Log10 Copies/mL
  Baseline | 2.28 (1.43) [62.1 to 73.5]
  48 weeks | 1.50 (0.45)

7. Secondary Outcome: Change From Baseline in CD4+ T-cell Counts in Aging Participants After 48 Weeks of Raltegravir Treatment
Description: Mean CD4+ T-cell counts were determined in aging participants (>=50 years old at initiation of raltegravir treatment) at baseline and after 48 weeks of raltegravir treatment was determined. A positive change from baseline indicates an increase in CD4+ T-cell count.
Time Frame: Baseline and 48 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: CD4+ T-cells/µL
Arm/Group | Aging Participants
Number analyzed (Participants) | 227
CD4+ T-cells/µL
  Baseline | 534.4 (297.48) [37.7 to 88.6]
  Change from Baseline at 48 weeks: n=202 | 63.2 (183.43)

8. Secondary Outcome: Change From Baseline in Mean Framingham Risk Score for the 10-Year Cardiovascular Risk in Aging Participants After 48 Weeks of Raltegravir Treatment
Description: Mean Framingham Risk for 10-year cardiovascular risk was determined in aging participants (>=50 years old at initiation of raltegravir treatment). Points were allotted for each of following 8 risk factors : sex, age, systolic blood pressure, treatment for hypertension, smoking, diabetes, total cholesterol, and high-density lipoprotein. The sum of the points for each participant was assigned a percent 10-year cardiovascular risk on a lookup table, and could range from 0% to 100%. The mean Framingham Risk for 10-year cardiovascular risk was then calculated for the analysis population. The change from baseline was calculated as Baseline minus Week 48; a positive change indicates reduced risk. This Outcome Measure was added with Amendment 1 and applies only to aging participants.
Time Frame: Baseline and 48 weeks
Population: The analysis set included aging participants (Prolonged Participants and Newly Enrolled Participants) who received at least one dose of raltegravir during the observation period and had evaluable results.
Measure: Mean (Standard Deviation); unit: Percentage risk
Arm/Group | Aging Participants
Number analyzed (Participants) | 105
Percentage risk
  Score at Baseline | 24.1 (17.5) [37.7 to 88.6]
  Change from Baseline at 48 weeks: n=65 | 1.1 (10.9)

9. Secondary Outcome: Change From Baseline in Mean D:A:D Risk Score for the 5-Year Cardiovascular Risk in Aging Participants After 48 Weeks of Raltegravir Treatment
Description: Mean Data Collection on Adverse Events of Anti-HIV Drugs (D:A:D) Risk Score for 5-year cardiovascular risk was determined in aging participants (>=50 years old at initiation of raltegravir treatment) at Baseline and after 48 weeks of raltegravir treatment. The score included the following 8 risk factors: sex, age, systolic blood pressure, family cardiovascular disease history, current smoking, previous cigarette smoker, diabetes, total cholesterol, high-density lipoprotein, currently on indinavir, currently on lopinavir, currently on abacavir, duration and current use of indinavir and duration and current use of lopinavir. The D:A:D Risk Score is interpreted as low: <1%; moderate: 1-5%; high: 5-10%; and very high: >10%. The change from baseline was calculated as Week 48 minus Baseline; a positive change indicates increased risk. This Outcome Measure was added with Amendment 1 and applies only to aging participants.
Time Frame: Baseline and 48 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage risk
Arm/Group | Aging Participants
Number analyzed (Participants) | 91
Percentage risk
  Score at Baseline | 9.4 (8.7) [37.7 to 88.6]
  Change from Baseline at 48 weeks: n=57 | 4.2 (9.5)

10. Secondary Outcome: Percentage of Aging Participants With Concomitant Diseases at Baseline
Description: The percentage of aging participants with Baseline comorbidities was reported. This Outcome Measure was added with Amendment 1 and applies only to aging participants.
Time Frame: Baseline
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Aging Participants
Number analyzed (Participants) | 227
Percentage of participants | 93.8

11. Secondary Outcome: Percentage of Aging Participants Taking Concomitant Medications at Baseline
Description: The percentage of aging participants taking concomitant medication in addition to their other antiretroviral therapy was reported. This Outcome Measure was added with Amendment 1 and applies only to aging participants.
Time Frame: Baseline
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Aging Participants
Number analyzed (Participants) | 227
Percentage of participants | 74.9

ADVERSE EVENTS:
Time Frame: Overall Participants: up to 48 weeks; Initial Cohort Participants: up to 96 weeks; Aging Participants: up to 48 weeks.
Description: Overall Participants and Aging Participants: MedDRA version 17.1; Initial Cohort Participants: MedDRA version 14.1.
Groups:
- Initial Cohort Participants: HIV-1 infected participants received raltegravir 400 mg tablet orally twice daily for 96 weeks in combination with other antiretroviral drugs under conditions representative of standard of clinical practice for HIV-1 patients in Germany.
Arm/Group | Overall Participants | Initial Cohort Participants | Aging Participants
Serious Adverse Events (participants affected / at risk) | 34/451 | 25/272 | 17/227
Other Adverse Events (participants affected / at risk) | 0/451 | 0/272 | 0/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Participants (N=451) | Initial Cohort Participants (N=272) | Aging Participants (N=227)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (2) | 0 (0) | 1 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Spirochaetal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (2) | 0 (0) | 1 (2)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram Q wave abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 2 (2) | 2 (2)
Transaminases increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1)
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study will be published by the sponsor according to the current guidelines for publication. The Contract Research Organization will assist the sponsor with initial publication. Further details will be laid down in the financial agreement between the sponsor and the Contract Research Organization.